CLINICAL TRIAL: NCT07068477
Title: Values Assessment Tailored for Women With Metastatic Breast Cancer and Their Caregivers: Adaptation and Pilot Study of a Values Assessment Tool (VAsT)
Brief Title: Adaptation of a Values Assessment Tool
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: LCCC2201
Record Dates: First submitted 2025-06-26; First posted 2025-07-16 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Cancer; Metastatic Breast Cancer
Keywords: African American; Latinx; Alaskan Native; Short Graphic Values History
MeSH Terms: conditions — Neoplasms; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Values assessment tool (Experimental): Participants are assessed at baseline and every clinic visit for 3 months
  Interventions: Behavioral: Values Assessment Tool

INTERVENTIONS:
Behavioral: Values Assessment Tool — The Values Assessment Tool was provided to the participants at baseline and every clinic visit for 3 months

SUMMARY:
The primary purpose of this study is to evaluate the effect of values assessment tool on patient and caregiver perception of decisional conflict, and communication with their oncology clinician.

DETAILED DESCRIPTION:
Incorporating patient values into shared decision-making is essential for individuals diagnosed with metastatic cancer. This is especially critical for women who identify as Black/African American, Latinx/Hispanic, or American Indian/Alaskan Native, as research indicates these groups face a higher risk of poor prognostic communication, worse health outcomes, and increased likelihood of metastatic cancer diagnoses compared to non-Hispanic White adults.

Black/African American women in the South, including North Carolina, experience the highest breast cancer mortality rates in the United States. In North Carolina, the majority of women diagnosed with metastatic breast cancer (mBC) are either non-Hispanic White (159 per 100,000) or Black/African American (164 per 100,000). This study aims to ensure that at least 40% of participants are Black/African American women.

While the Short Graphic Values History (SGVH) tool has been used in general ambulatory care, it has not been tested or adapted for use in cancer care settings. Based on interviews with individuals living with mBC and their care partners, a new Values Assessment Tool (VAsT) has been developed for integration into cancer care.

This single-arm prospective study will enroll 40 women with mBC and their caregivers. Baseline data will be collected at diagnosis, followed by deployment of the VAsT in clinic settings. Follow-up feedback will be obtained to assess real-world usability and relevance of the tool in supporting shared decision-making in cancer care.

ELIGIBILITY:
Inclusion Criteria

1. Age ≥18 years
2. Diagnosed with metastatic breast cancer.
3. Understand and read English.
4. Receive care or anticipate receiving care at the North Carolina Cancer Hospital ambulatory cancer clinic or affiliated community cancer clinic.
5. Able to understand and participate in study procedures for length of study.

Exclusion Criteria

1. All subjects meeting any of the exclusion criteria at baseline will be excluded from study participation:
2. Unable to provide consent, unable to communicate verbally.
3. Unable to understand or read English.
4. Enrolled in hospice care.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2023-01-05 (Actual); Primary Completion 2026-08-24 (Estimated); Study Completion 2026-08-24 (Estimated)

PRIMARY OUTCOMES:
Decisional engagement | Baseline and every clinic visit for 3 months
  Values Assessment Tool participants will be assessed using decisional engagement, Patient-Centered Communication in Cancer Care (PCC-Ca) 36.
  Each item included in the PCC-Ca instrument consists of a question stem and five response options. The response options are scored from 1 to 5, with higher scores representing better communication; for example, where 1 = Never and 5 = Always. There are no reverse-scored items. Some items have a sixth "does not apply" option. This response is not scored.
Decisional conflict | Baseline and every clinic visit for 3 months
  Decisional Conflict will be assessed using the Decisional Conflict Scale (10-item low literacy version).
  Scoring and Interpretation: Items are given a score value of: 0 = 'yes'; 2 = 'unsure'; 4 = 'no'
  Total Score: 10 items [items 1-10 inclusive] are: a) summed; b) divided by 10; and c) multiplied by 25.
  Scores range from 0 [no decisional conflict] to 100 [extremely high decisional conflict]
Communication perceptions | Baseline and every clinic visit for 3 months
  Communication perceptions will be assessed using Patient-Centered Communication in Cancer Care (PCC-Ca) 36.
  Each item included in the PCC-Ca instrument consists of a question stem and five response options. The response options are scored from 1 to 5, with higher scores representing better communication; for example, where 1 = Never and 5 = Always. There are no reverse-scored items. Some items have a sixth "does not apply" option. This response is not scored.

SECONDARY OUTCOMES:
The number of participants who started and completed | Baseline and 3 months
  The number of participants who started and completed using the Values Assessment Tool will be presented.
Shared decision making evaluation | Baseline and 3 months
  Shared decision-making will be evaluated through a combination of qualitative semi-structured interviews and audio recordings of clinical encounters with enrolled patient participants, conducted both before and after the use of the Short Graphic Values History (SGVH) tools.
  Open-ended feedback from participants will undergo content analysis to identify key themes. These insights will be used to prioritize recommendations for refining the next iteration of the SGVH tool intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Lorinda Coombs, PhD, FNP-BC, AOCNP, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- UNC Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials